CLINICAL TRIAL: NCT02741726
Title: Effect of Combined-acupoint or Single-acupoint Stimulation Before Surgery on Post Mastectomy Pain: a Multicentre Randomised Controlled Trial
Brief Title: Analgesia by Single or Dual Acupoints Stimulation After Radical Mastectomy
Acronym: ASDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Doctor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJH-A-2016-04-12
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- dual acupoint stimulation (Experimental): The acupoints of dual point group are bilateral Neiguan points(PC6) combined with Danzhong point(RN17), electric stimulation was given through electrode attached to the acupoints.
  Interventions: Device: acupoint stimulation
- single acupoint stimulation (Experimental): The acupoints of single point group is bilateral Neiguan points(PC6), Electric stimulation was given through electrode attached to the acupoints.
  Interventions: Device: acupoint stimulation
- no stimulation (Placebo Comparator): false stimulation group only attach electrodes without electric current.
  Interventions: Device: no stimulation

INTERVENTIONS:
Device: acupoint stimulation — Electric stimulation was given through electrode attached to acupoints
  Other Names: transcutaneous electrical acupoint stimulation
  Arms: dual acupoint stimulation; single acupoint stimulation
Device: no stimulation — patients were only attached electrodes without electric current
  Arms: no stimulation

SUMMARY:
The purpose of this study is to compare the effects of dual acupoints and single acupoint transcutaneous electrical acupoint stimulation (TEAS) pretreatment on incidence of Post-Mastectomy Pain Syndrome(PMPS) in patients undergoing operation of breast cancer.

DETAILED DESCRIPTION:
Patients were randomly assigned to three groups, receiving 30min TEAS before anesthesia respectively. The acupoints of dual point group are bilateral Neiguan points(PC6) combined with Danzhong point(RN17), single point group is bilateral Neiguan points(PC6), and the false stimulation group only attach electrodes without electric current. The frequency of TEAS is set to 2/15 Hz. Intraoperative anesthetic dosage of propofol and remifentanil was recorded. Three and six months after surgery, follow-up about chronic pain was made by telephone or face-to-face using the follow-up questionnaire. The adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for operation of breast cancer；
* ASA（American Society of Anesthesiologists）I-II；
* Aged between 18 and 65；
* Informed consented。

Exclusion Criteria:

* Suffered from the contraindication of TEAS including the local skin breakage, infection or planted with the electrophysiology device；
* Unable to communicate and coordinate with the researcher, such as suffering from language comprehension deficits or mental diseases；
* Certain/suspicious addiction with alcohol, analgesics or other drugs；
* Unstable Angina or myocardial infarction occurred in 3 months; NYHA（New York Heart Association） is 3 or higher;
* Blood pressure ≥ 180/110 mm Hg while preoperative visiting;
* Suffered from diabetic complications including diabetic ketoacidosis, hyperosmolar coma, infection, macroangiopathy, diabetic nephropathy, retinopathy, cardiomyopathy, neuropathy and diabetic foot;
* Severe dysfunction of liver or kidney meaning one of ALT（Alanine Transaminase）, AST（Aspartate Transaminase）, ALP（alkaline phosphatase） or TBIL（total bilirubin） is 2 times higher that normal or creatinine clearance < 30 ml/min or serum creatinine > 177umol/L;
* Participate in the other clinical trial 3 month before the enrollment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic pain six months after surgery | six months after surgery

SECONDARY OUTCOMES:
Incidence of chronic pain three months after surgery | three months after surgery
Remifentanil consumption during the surgery | from start of surgery to end of surgery, at an average of 2.5 hours
the time to the first verbal response | end of the anesthetics infusion to patient's first response to verbal command,on an average of 30 minutes
the time to extubation | end of the anesthetics infusion to extubation,on an average of 30 minutes
postoperative nausea and vomiting within 24 h after surgery | end of surgery to 24 hours after surgery,on an average of 24 hours
respiratory depression within 24 hours after surgery | end of surgery to 24 hours after surgery,on an average of 24 hours
patients' s satisfaction scores on analgesia within 24 hours after surgery | end of surgery to 24 hours after surgery,on an average of 24 hours
Visual Analogue Scale scores within 24 hours after surgery | end of surgery to 24 hours after surgery,on an average of 24 hours
demand of rescue analgesics within 24 hours after surgery | end of surgery to 24 hours after surgery,on an average of 24 hours
pain score at 3m after surgery | three months after surgery
pain score at 6m after surgery | six months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Study Chair — Air Force Military Medical University, China
Locations (6):
- China (6):
  - First Afiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - People's hospital of Zhengzhou University, Zhengzhou, Henan
  - First Afiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tangdu Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - First Afiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
IPD including those about primary endpoint and secondary endpoints would be available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the data will become available after manuscript published, for 5 years.

REFERENCES:
- [Derived] Lu Z, Wang Q, Sun X, Zhang W, Min S, Zhang J, Zhao W, Jiang J, Wang Y, Zhu Y, Zheng L, Wang Y, Guo Y, Zhang L, Wang L, Lei C, Liu T, Yang X, Zhang J, Li C, Zhang N, Dong H, Xiong L. Transcutaneous electrical acupoint stimulation before surgery reduces chronic pain after mastectomy: A randomized clinical trial. J Clin Anesth. 2021 Nov;74:110453. doi: 10.1016/j.jclinane.2021.110453. Epub 2021 Jul 13. PMID 34271271